CLINICAL TRIAL: NCT01645072
Title: Efficacy of Low Glycemic Index Diet Therapy in Children With Refractory Epilepsy - A Randomized Controlled Trial
Brief Title: Low Glycemic Index Diet Therapy in Children With Refractory Epilepsy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sheffali Gulati, Additional Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIIMS
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Refractory Epilepsy
Keywords: Drug refractory epilepsy; Dietary therapy; ketogenic diet; childhood epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low glycemic index diet (Experimental): The patients will be started on low glycemic index diet.
  Interventions: Other: Low glycemic index diet
- Control group (Other): Standard care. The control group will receive their usual diet without any alteration. No changes will be made to the patients' antiepileptic medication during the 4-week baseline or the 3-month study periods in both the intervention and control groups, unless medically indicated; e.g. drug side effects, or status epilepticus; in which case appropriate changes will be made to their medications and same will be documented.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Low glycemic index diet — Diet modification in addition to ongoing anti epileptic drug treatment. Medium and high-GI carbohydrates (GI >55) will be eliminated from the diet and only food items with low glycemic index (GI <55) will be allowed. Parent will be given a list of low glycemic index food items. They will also be given a list of food items (medium and high glycemic index) which should be avoided.
  Arms: Low glycemic index diet
Other: Control group — The ongoing anti epileptic drug treatment will be continued without change.
  Arms: Control group

SUMMARY:
Epilepsy is a frequent cause of morbidity in the pediatric age group. Many catastrophic epilepsies present during infancy and childhood1. Seizures in these epileptic disorders are difficult to control; sometimes only at the expense of multiple and toxic levels of antiepileptic medications. The shortcomings of antiepileptic drug therapy and epilepsy surgery warrants the need for alternative treatments. Ketogenic diet is effective for refractory epilepsies (33% of patients with refractory epilepsy have more than 50% reduction in seizures from the baseline and 15-20% become seizure free) and has gained widespread acceptance. Low glycemic index diet treatment (LGIT) is designed as a variant of ketogenic diet. There are retrospective studies on LGIT in childhood refractory epilepsy reporting seizure reduction comparable to that of patients on ketogenic diet. There have been no randomized controlled trials assessing the efficacy of the low glycemic index diet in refractory epilepsy. In this study we plan to assess the efficacy of LGIT among children with drug refractory epilepsy.

DETAILED DESCRIPTION:
Each patient will undergo detailed clinical evaluation according to a structured proforma. Seizure type, frequency, age at onset, perinatal details, family history, developmental status and treatment history will be recorded. Corticosteroids or ACTH (if patient is already on) would be tapered off 2 weeks before starting LGIT. All co-medications will be changed to carbohydrate free preparations, wherever available only in the intervention group.

Eligible patients will be randomized in to two groups: the intervention and the control arm. Both groups will undergo a baseline four week observation period, during which parents will be asked to maintain a daily seizure log; recording seizure type, duration and frequency. In the intervention arm, the children will be started on low glycemic index diet after this 4-week baseline period. The control group will receive their usual diet without any alteration. No changes will be made to the patients' antiepileptic medication during the 4-week baseline or the 3-month study periods in both the intervention and control groups, unless medically indicated; e.g. drug side effects, or status epilepticus; in which case appropriate changes will be made to their medications and same will be documented. The drop out from the intervention group will be documented along with the reason for the same. At the end of the 3 month study period patient in the intervention arm will be continued with the LGIT but that will not come under the purview of this study. At the end of three months study period, patients in the control arm will be offered the option of low glycemic index diet treatment.

Low glycemic index diet administration

1. Three day food intake by recall method will be documented
2. The calorie requirement would be calculated as per the recommended daily allowance (RDA) for the ideal weight for that age
3. Diet regime will be explained to the parents
4. Patients (wherever applicable) and their parents will be given diet counseling
5. LGIT will be started on out patient basis.
6. Medium and high-GI carbohydrates (GI >55) will be eliminated from the diet and only food items with low glycemic index (GI <55) will be allowed. Parent will be given a list of low glycemic index food items33. They will also be given a list of food items (medium and high glycemic index) which should be avoided. (Appendix)
7. Total carbohydrates intake will be restricted to 10% of caloric intake/ day (maximum 40-60 g/day).
8. Carbohydrate values of various food items will be explained in detail, and carbohydrate exchange lists will be provided to the parent. Three to four 15 gram carbohydrate exchanges will be allowed in a day. (Appendix)
9. Fats (e.g. cream, butter, oils and ghee) can be taken by the patient without any restriction.
10. Proteins intake will be allowed up to 30% of the total caloric intake per day (cheese, fish, eggs, chicken and soya products).
11. Sample menu will be discussed with the parent.
12. Clear carbohydrate free fluids will not be restricted.

Follow up Children will be reviewed as outpatients at 1, 2 and 3 months. A three day dietary intake chart will be reviewed at each visit to compute calorie and carbohydrate intake, and to evaluate and reinforce compliance with the prescribed diet. Weight will be checked at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 2 -15 years with refractory epilepsy*
2. Willing to come for regular follow up
3. No motivational or psychosocial issues in the family which would preclude compliance with the diet * Refractory epilepsy is defined as seizures persisting daily or more than 7 per week despite the adequate trials of at least three tolerated and appropriately chosen anti-epileptic drugs including one newer antiepileptic drug (either alone or in combination). In case of infantile spasms, epileptic spasms with the onset before 2 years of age, with or without electroencephalographic evidence of hypsarrhythmia or its variants, persisting for more than 3 weeks, at least 7 cluster per week, despite treatment with at least 2 appropriate AEDs, and any one of the following; corticosteroids or vigabatrin will be considered as eligible for inclusion.

Exclusion Criteria:

1. Surgically remediable cause for refractory epilepsy
2. Suspected mitochondrial disorder or diagnosed with a disorder in which high fat diet is contraindicated
3. Previously received ketogenic diet or modified Atkins diet
4. Chronic systemic disease like chronic kidney disease, chronic liver disease, heart disease (congenital and acquired) and chronic respiratory illness

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-08 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Seizure control | 3 months
  Proportion of patients who achieve > 50% seizure reduction (Seizure frequency measured as average seizure per week in the preceding 4 week period) from the baseline

SECONDARY OUTCOMES:
Adverse events | 3 months
  Proportion and nature of adverse events in both the groups
Withdrawal rate | 3 months.
  Proportion of patients withdrawing from the LGIT plus antiepileptic drug treatment group during the study period and reasons for withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Sheffali Gulati, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India